CLINICAL TRIAL: NCT04208412
Title: A Randomized, Double-blind, Placebo-controlled, Phase II, Cross-over Clinical Trial Evaluating the Efficacy and Safety of KVD900, an Oral Plasma Kallikrein Inhibitor, in the On-demand Treatment of Angioedema Attacks in Adult Subjects With Hereditary Angioedema Type I or II
Brief Title: A Phase II, Cross-over Clinical Trial Evaluating the Efficacy and Safety of KVD900 (Sebetralstat) in the On-demand Treatment of Angioedema Attacks in Adult Subjects With Hereditary Angioedema Type I or II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KVD900-201
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Angioedema
Keywords: Sebetralstat
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Subjects received a single dose of 600 mg KVD900.
  Interventions: Drug: KVD900
- Part 2 - Sequence 1: 600 mg KVD900, Then Placebo (Experimental): Subjects received a single dose of 600 mg KVD900 to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of placebo to treat the second eligible HAE attack.
  Interventions: Drug: KVD900; Other: Placebo
- Part 2 - Sequence 2: Placebo, Then 600 mg KVD900 (Experimental): Subjects received a single dose of placebo to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of 600 mg KVD900 to treat the second eligible HAE attack.
  Interventions: Drug: KVD900; Other: Placebo

INTERVENTIONS:
Drug: KVD900 — KVD900 tablet 600 mg
Other: Placebo — KVD900-matched Placebo Tablet
  Arms: Part 2 - Sequence 1: 600 mg KVD900, Then Placebo; Part 2 - Sequence 2: Placebo, Then 600 mg KVD900

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, phase II, cross-over clinical trial evaluating the efficacy and safety of KVD900, in the treatment of hereditary angioedema attacks in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult subjects 18 years of age and older.
* Confirmed diagnosis of HAE type I or II at anytime in the medical history
* At least 3 documented HAE attacks in the past 93 days, as supported by medical history.
* Access to and ability to use conventional attack treatment for attacks of HAE
* Adequate organ functions
* Females of childbearing potential must agree to use highly effective birth control from the Screening visit until the end of the trial follow-up procedures.
* Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months, do not require contraception during the study
* Males with female partners of childbearing potential must agree to be abstinent or else use a highly effective method of birth control as defined in inclusion 6 from the Screening visit until the end of the trial follow-up procedures
* Provide signed informed consent and are willing and capable of complying with study requirements and procedures

Exclusion Criteria:

* Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1 inhibitor (C1-INH) deficiency, HAE with normal C1-INH (also known as HAE type III), idiopathic angioedema, or angioedema associated with urticaria
* Current use of C1INH, androgens, or tranexamic acid for HAE prophylaxis
* Use of angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications with systemic absorption (such as oral contraceptives or hormonal replacement therapy) within 93 days prior to initial study treatment.
* Use of androgens (e.g. stanozolol, danazol, oxandrolone, methyltestosterone, testosterone) or antifibrinolytics within 30 days prior to initial study treatment.
* Use of lanadelumab within 10 weeks prior to initial study treatment.
* Use of strong CYP3A4/CYP2C9 inhibitors and inducers during participation in the trial
* Clinically significant abnormal ECG at Visit 1 and pre-dose at Visit 2. This includes, but is not limited to, a QT interval by Fredericia, QTcF > 470 msec (for women) or > 450 msec (for men), a PR > 220 msec or ventricular and/or atrial premature contractions that are more frequent than occasional and/or occur as couplets or higher in grouping
* Any clinically significant history of angina, myocardial infarction, syncope, clinically significant cardiac arrhythmias, left ventricular hypertrophy, cardiomyopathy, or any other cardiovascular abnormality
* Any other systemic dysfunction (e.g., gastrointestinal, renal, respiratory, cardiovascular) or significant disease or disorder which, in the opinion of the Investigator, would jeopardize the safety of the subject by taking part in the trial
* History of substance abuse or dependence that would interfere with the completion of the study, as determined by the Investigator
* Known lactose allergy or intolerance
* Known hypersensitivity to KVD900 or placebo or to any of the excipients
* Participation in an interventional investigational clinical study within 93 days or within 5 half-lives of the last dosing of investigational drug (whichever is longer) prior to initial study treatment
* Any pregnant or breast-feeding subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals, Ltd.
Locations (25):
- United States (6):
  - KalVista Investigative Site, Scottsdale, Arizona
  - KalVista Investigative Site, Centennial, Colorado
  - KalVista Investigative Site, Chevy Chase, Maryland
  - KalVista Investigative Site, Cincinnati, Ohio
  - KalVista Investigative Site, Dallas, Texas
  - KalVista Investigative Site, Spokane, Washington
- KalVista Investigative Site, Vienna, Austria
- Czechia (3):
  - KalVista Investigative Site, Brno
  - KalVista Investigative Site, Hradec Králové
  - KalVista Investigative Site, Pilsen
- Germany (3):
  - KalVista Investigative Site, Berlin
  - KalVista Investigative Site, Frankfurt
  - KalVista Investigative Site, Mörfelden-Walldorf
- KalVista Investigative Site, Budapest, Hungary
- Italy (3):
  - KalVista Investigative Site, Milan
  - KalVista Investigative Site, Milano-2
  - KalVista Investigative Site, Padua
- KalVista Investigative Site, Amsterdam, Netherlands
- KalVista Investigative Site, Skopje, North Macedonia
- Poland (2):
  - KalVista Investigative Site, Krakow
  - KalVista Investigative Site, Warsaw
- United Kingdom (4):
  - KalVista Investigative Site, Camberley
  - KalVista Investigative Site, Cambridge
  - KalVista Investigative Site, London
  - KalVista Investigative Site, Newcastle

REFERENCES:
- [Derived] Aygoren-Pursun E, Zanichelli A, Cohn DM, Cancian M, Hakl R, Kinaciyan T, Magerl M, Martinez-Saguer I, Stobiecki M, Farkas H, Kiani-Alikhan S, Grivcheva-Panovska V, Bernstein JA, Li HH, Longhurst HJ, Audhya PK, Smith MD, Yea CM, Maetzel A, Lee DK, Feener EP, Gower R, Lumry WR, Banerji A, Riedl MA, Maurer M. An investigational oral plasma kallikrein inhibitor for on-demand treatment of hereditary angioedema: a two-part, randomised, double-blind, placebo-controlled, crossover phase 2 trial. Lancet. 2023 Feb 11;401(10375):458-469. doi: 10.1016/S0140-6736(22)02406-0. PMID 36774155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 84 subjects were enrolled, of which 16 were screen failures. The majority of screen failures were due to inclusion criterion not met.
Pre-assignment Details: A total of 68 subjects were entered into the open-label safety, tolerability and PK section (Part 1) and subsequently into Part 2, where all 68 subjects were randomized, with 34 subjects randomized to Sequence 1 (600 mg KVD900; Placebo) and 34 subjects randomized to Sequence 2 (Placebo; 600 mg KVD900).
Groups:
- 600 mg KVD900, Then Placebo: Subjects received a single dose of 600 mg KVD900 to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of placebo to treat the second eligible HAE attack.
- Placebo, Then 600 mg KVD900: Subjects received a single dose of placebo to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of 600 mg KVD900 to treat the second eligible HAE attack.
Period: Overall Study
Arm/Group | 600 mg KVD900, Then Placebo | Placebo, Then 600 mg KVD900
Started | 34 | 34
Completed | 25 | 28
Not Completed | 9 | 6
Not completed — Early discontinuation per protocol; sufficient number of subjects completed the study | 8 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 mg KVD900, Then Placebo | Placebo, Then 600 mg KVD900 | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.97) | 35.5 (13.12) | 38.3 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 12 | 19 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 34 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: meters] | 1.711 (0.0837) | 1.730 (0.1039) | 1.720 (0.0941)
Weight [Mean (Standard Deviation); unit: kg] | 79.89 (18.335) | 82.04 (18.865) | 80.97 (18.495)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.242 (5.7344) | 27.336 (5.2691) | 27.289 (5.4656)

OUTCOME MEASURES:

1. Primary Outcome: Time to Conventional Attack Treatment Use Within 12 Hours of Study Drug (Full Analysis Set)
Description: The primary variable for statistical comparison between treatments in Part 2 of the study was time to use of conventional attack treatment (pdC1INH or rhC1INH intravenous [iv] or icatibant) within 12 hours of study drug.
  Censoring occurs where a subject did not use conventional attack treatment within 12h post-study drug dosing.
  When an endpoint result was non-calculable (NC) within 12 hours, if the event did occur, the event must have occurred >12 hours following study drug.
Time Frame: 12 hours
Population: A total of 53/68 subjects (77.9%) completed the study. First interquartile values and 95% CI are NA (9.5 to NDA) and 8.0 (3.8 to NA) for the 600 mg KVD900 and Placebo Arm/Groups respectively. Here NA is identical to the footnote.
Measure: Median (95% Confidence Interval); unit: Time (h)
Groups:
- 600 mg KVD900; Placebo: In Sequence 1, subjects received a single dose of 600 mg KVD900 to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of placebo to treat the second eligible HAE attack.
  In Sequence 2, subjects received a single dose of placebo to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of 600 mg KVD900 to treat the second eligible HAE attack.
Arm/Group | 600 mg KVD900 | Placebo
Number analyzed (Participants) | 53 | 53
Time (h) | NA [NA to NA] — NA represents non-calculable (NC), defined as not enough subjects used conventional attack treatment within 12 hour to complete descriptive statistics | NA [NA to NA] — NA represents non-calculable (NC), defined as not enough subjects used conventional attack treatment within 12 hour to complete descriptive statistics
Statistical Analysis 1: Comparison: 600 mg KVD900 vs Placebo; Test type: Superiority; p = 0.0010, Wilcoxon Test (Gehan's Generalized)

2. Secondary Outcome: Proportion of HAE Attacks That Worsen in Severity by One Level or More on the PGI-S or Require Conventional Attack Treatment Within 12 Hours of Study Drug (Full Analysis Set)
Description: The proportion of participant's HAE attacks to either worsen in attack severity on the PGI-S by one level or more or conventional attack treatment (pdC1INH or rhC1INH intravenous [iv] or icatibant) use are listed with censored observations flagged. Frequencies (n, %) of subjects experiencing a worsening on the PGI-S by one level or more or using conventional attack treatment and the number censored are presented. "Y" Row indicates "participants who experienced a worsening in severity, and the "N" Row indicates participants who did not.
Time Frame: 12 hours
Population: A total of 53/68 subjects (77.9%) completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 600 mg KVD900 | Placebo
Number analyzed (Participants) | 53 | 53
Participants
  Y | 11 | 24
  N | 42 | 29
Statistical Analysis 1: Comparison: 600 mg KVD900 vs Placebo; Test type: Superiority; p = 0.0045, Prescott's Test

3. Secondary Outcome: Time to Either Worsening in HAE Attack Severity by One Level or More on the PGI-S or to Conventional Attack Treatment Use Within 12 Hours of Study Drug (Full Analysis Set)
Description: HAE attack severity assessed using the Patient Global Impression of Severity scale (PGI-S).
  Censoring occurs where a subject did not worsen in severity or use conventional attack treatment (pdC1INH or rhC1INH intravenous [iv] or icatibant) within 12h post-study drug dosing.
  When an endpoint result was non-calculable (NC) within 12 hours, if the event did occur, the event must have occurred >12 hours following study drug.
Time Frame: 12 hours
Population: A total of 53/68 subjects (77.9%) completed the study. First interquartile values and 95% CI are NA (5.9 to NA) and 3.0 (2.0 to 6.0) for the 600 mg KVD900 and Placebo Arm/Groups respectively. Here NA is identical to the footnote.
Measure: Median (95% Confidence Interval); unit: Time (h)
Arm/Group | 600 mg KVD900 | Placebo
Number analyzed (Participants) | 53 | 53
Time (h) | NA [NA to NA] — NA represents non-calculable (NC), defined as not enough subjects used conventional attack treatment within 12 hour to complete descriptive statistics | NA [6.0 to NA] — NA represents non-calculable (NC), defined as not enough subjects used conventional attack treatment within 12 hour to complete descriptive statistics
Statistical Analysis 1: Comparison: 600 mg KVD900 vs Placebo; Gehan's Generalized Wilcoxon Test: 600 mg KVD900 vs Placebo; Test type: Superiority; p < 0.0001, Wilcoxon Test (Gehan's Generalized)

4. Secondary Outcome: Time to Symptom Relief Defined as HAE Attack Rated as "A Little Better" or Higher on the PGI-C for Two Consecutive Time Points Within 12 Hours of Study Drug (Full Analysis Set)
Description: Change in HAE attack severity assessed using the Patient Global Impression of Change 7-point transition question (PGI-C).
  Censoring occurs where an attack rating of "a little better" or higher for two consecutive time points does not occur or conventional attack treatment is used within 12h post-study drug dosing.
  When an endpoint result was non-calculable (NC) within 12 hours, if the event did occur, the event must have occurred >12 hours following study drug.
Time Frame: 12 hours
Population: A total of 53/68 subjects (77.9%) completed the study. First interquartile values and 95% CI are 0.6 (0.6 to 1.5) and 2.0 (0.6 to 4.0) for the 600 mg KVD900 and Placebo Arm/Groups respectively. Here NA is identical to the footnote.
Measure: Median (95% Confidence Interval); unit: Time (h)
Groups:
- 600 mg KVD90; Placebo: In Sequence 1, subjects received a single dose of 600 mg KVD900 to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of placebo to treat the second eligible HAE attack.
  In Sequence 2, subjects received a single dose of placebo to treat the first eligible HAE attack. Following resolution of this attack, subjects received a second single dose of 600 mg KVD900 to treat the second eligible HAE attack.
Arm/Group | 600 mg KVD90 | Placebo
Number analyzed (Participants) | 53 | 53
Time (h) | 1.6 [1.5 to 3.0] | 9.0 [4.0 to NA] — NA represents non-calculable (NC), defined as not enough subjects used conventional attack treatment within 12 hour to complete descriptive statistics
Statistical Analysis 1: Comparison: 600 mg KVD90 vs Placebo; Test type: Superiority; p < 0.0001, Wilcoxon Test (Gehan's Generalized)

5. Secondary Outcome: Time to Symptom Relief Defined as 50% Reduction in Composite VAS Score for Three Consecutive Time Points Within 12 Hours of Study Drug (Full Analysis Set)
Description: The HAE attack symptoms were assessed on a 100 mm visual analogue scale (VAS) ranging from 0 (none) to 100 (very severe).
  The Composite VAS score is defined as the mean score across all symptoms. Censoring occurs where a ≥50% reduction in Composite VAS Score for three consecutive time points does not occur or conventional attack treatment is used within 12h post-study drug dosing.
  When an endpoint result was non-calculable (NC) within 12 hours, if the event did occur the event must have occurred >12 hours following study drug.
Time Frame: 12 hours
Population: A total of 53/68 subjects (77.9%) completed the study. First interquartile values and 95% CI are 2.5 (1.5 to 3.5) and 6.0 (3.0 to NA) for the 600 mg KVD900 and Placebo Arm/Groups respectively. Here NA is identical to the footnote.
Measure: Median (95% Confidence Interval); unit: Time (h)
Arm/Group | 600 mg KVD900 | Placebo
Number analyzed (Participants) | 53 | 53
Time (h) | 6.0 [3.0 to 9.0] | NA [NA to NA] — NA represents non-calculable (NC), defined as not enough subjects used conventional attack treatment within 12 hour to complete descriptive statistics
Statistical Analysis 1: Comparison: 600 mg KVD900 vs Placebo; Test type: Superiority; p < 0.0001, Wilcoxon Test (Gehan's Generalized)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the maximum duration of randomized subject participation from screening until final visit (up to 19 weeks).
Description: Safety was evaluated for Parts 1 and 2 by the following:
  * AEs, including serious adverse events (SAEs).
  * Laboratory test results (clinical chemistry, hematology, coagulation, and urinalysis).
  * Vital signs (systolic blood pressure [SBP], diastolic blood pressure [DBP], pulse rate, respiratory rate and body temperature).
  * Physical exam findings.
  * ECG results.
  * Pregnancy test (female subjects of child-bearing potential)
Groups:
- Part 1: 600 mg KVD900: Subjects received a single dose of 600 mg KVD900.
- Part 2: 600 mg KVD900: Subjects received a single dose of 600 mg KVD900 to treat eligible HAE attack.
- Part 2: Placebo: Subjects received a single dose of placebo to treat eligible HAE attack.
Arm/Group | Part 1: 600 mg KVD900 | Part 2: 600 mg KVD900 | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/58 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/58 | 0/55
Other Adverse Events (participants affected / at risk) | 7/68 | 8/58 | 5/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: 600 mg KVD900 (N=68) | Part 2: 600 mg KVD900 (N=58) | Part 2: Placebo (N=55)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT04208412/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04208412/SAP_001.pdf